CLINICAL TRIAL: NCT04651309
Title: Assessment of Labour Progress by Intrapartum Ultrasound: Can it Reduce the Incidence of Chorioamnionitis?
Brief Title: Assessment of Labour Progress by Intrapartum Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0118-17-KMC
Record Dates: First submitted 2020-11-15; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Pregnancy Related; Fever; Chorioamnionitis; Labor Complication
MeSH Terms: conditions — Fever; Chorioamnionitis; Obstetric Labor Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Other): Labor progress assessed by US, avoiding digital exams as much as possible;
  Interventions: Other: Transperineal Ultrasound
- Control group (No Intervention): Labor progress assessed according to the regular protocol

INTERVENTIONS:
Other: Transperineal Ultrasound — The ultrasound examination will be conducted using the technique described by Hassan et al (2013). Briefly, transperineal ultrasound images are obtained by placing a covered transducer between the labia below the symphysis pubis. Small lateral movements of the probe are then made to align the ultrasound beam in a midsagittal orientation to include the whole cervical length after which the probe is rotated 90 degrees in order to measure the cervical dilatation. The probe is rotated up and down until the echogenic circle of the cervix is seen. Please note that this technique is widely used within the delivery room and that the ultrasound machine that will be used is frequently used within the delivery room.
  Arms: Ultrasound group

SUMMARY:
Assessment of labor progress via digital exams is considered the standard of care in most delivery rooms. However, this method can be stressful, painful and imprecise and multiple exams increase the risk for chorioamnionitis. Trans-perineal ultrasound (TPUS) was found to be an objective noninvasive way to monitor labor progress. The study aim is to investigate whether, in nulliparous women, the use of TPUS during labor can reduce the number of vaginal exams and the incidence of chorioamnionitis.

DETAILED DESCRIPTION:
The prevalence of chorioamnionitis in term deliveries is 1-5% and in preterm deliveries the numbers can be as high as 25%. Most infections are a result of an ascending infection of the normal vaginal flora. Among risk factors are nulliparity, rupture of membranes, an extended duration of labor, multiple vaginal examinations and GBS colonization.

The digital vaginal examination remains to this day the standard method for evaluating the patient's cervical status. However, this method is both highly subjective as well as painful and stressogenic for the patients.

In recent years there has been great progress in the field of translabial/transperineal sonography. There have been several studies which showed that this technique could be as useful as digital examinations in helping clinicians predict the course of labor. Recent studies demonstrate that using transperineal sonography can reduce the perception of pain compared with routine digital vaginal examinations. Even so, there has been little evidence as to whether using perineal ultrasound may also reduce peripartum and puerperal infections and if using sonography and refraining from digital examinations affects the course and duration of labor.

Our objective is to evaluate whether the incidence of chorioamnionitis or fever can be decreased. This goal would hopefully be achieved by assessing the progression of labor using mostly transperineal ultrasound, thus avoiding digital vaginal examination as much as possible.

The study would focus on primigravid women as they are known to be in a higher risk for infection and also other potential risk factors such as GBS carriers and PROM.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida
* Gestational age ≥ 37 weeks (according to 1st trimester sonography)
* Single fetus •Cephalic presentation

Exclusion Criteria:

o Other known active infection (such as URTI, UTI)

* Women who are taking immunosuppressive therapy
* Women who arrived in active labor and delivered before being assessed by a physician.
* Women with contra-indications for vaginal birth

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Fever and infection rates in each of the study arms | From admission to hospital for labor until 2 week post-partum
  Intrapartum and post partum fever rates will be evaluated in both the study and the control groups.
Number of digital exams in each of the study arms | From admission to hospital until delivery
  The number of digital exams will be counted in each of the study arms

CONTACTS AND LOCATIONS:
Overall Officials: Maya Oberman, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Maya Oberman, Rehovot, Israel

REFERENCES:
- [Background] Gabbe, Steven G, Obstetrics: normal and problem pregnancies , Seventh edition. ..2017
- [Background] Seaward PG, Hannah ME, Myhr TL, Farine D, Ohlsson A, Wang EE, Haque K, Weston JA, Hewson SA, Ohel G, Hodnett ED. International Multicentre Term Prelabor Rupture of Membranes Study: evaluation of predictors of clinical chorioamnionitis and postpartum fever in patients with prelabor rupture of membranes at term. Am J Obstet Gynecol. 1997 Nov;177(5):1024-9. doi: 10.1016/s0002-9378(97)70007-3. PMID 9396886
- [Background] Benediktsdottir S, Eggebo TM, Salvesen KA. Agreement between transperineal ultrasound measurements and digital examinations of cervical dilatation during labor. BMC Pregnancy Childbirth. 2015 Oct 24;15:273. doi: 10.1186/s12884-015-0704-z. PMID 26496894
- [Background] Yuce T, Kalafat E, Koc A. Transperineal ultrasonography for labor management: accuracy and reliability. Acta Obstet Gynecol Scand. 2015 Jul;94(7):760-765. doi: 10.1111/aogs.12649. Epub 2015 May 5. PMID 25846302
- [Background] Hassan WA, Eggebo T, Ferguson M, Gillett A, Studd J, Pasupathy D, Lees CC. The sonopartogram: a novel method for recording progress of labor by ultrasound. Ultrasound Obstet Gynecol. 2014 Feb;43(2):189-94. doi: 10.1002/uog.13212. PMID 24105734
- [Background] Seval MM, Yuce T, Kalafat E, Duman B, Aker SS, Kumbasar H, Koc A. Comparison of effects of digital vaginal examination with transperineal ultrasound during labor on pain and anxiety levels: a randomized controlled trial. Ultrasound Obstet Gynecol. 2016 Dec;48(6):695-700. doi: 10.1002/uog.15994. Epub 2016 Nov 8. PMID 27300158
- [Derived] Oberman M, Avrahami I, Lavi Shoseyov N, Kandel A, Ben-Arie A, Sacagiu M, Vaisbuch E, Levy R. Assessment of labor progress by ultrasound vs manual examination: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Feb;5(2):100817. doi: 10.1016/j.ajogmf.2022.100817. Epub 2022 Nov 16. PMID 36400420
- [Derived] Hsu S, Selen DJ, James K, Li S, Camargo CA Jr, Kaimal A, Powe CE. Assessment of the Validity of Administrative Data for Gestational Diabetes Ascertainment. Am J Obstet Gynecol MFM. 2023 Feb;5(2):100814. doi: 10.1016/j.ajogmf.2022.100814. Epub 2022 Nov 15. PMID 36396038